CLINICAL TRIAL: NCT05873751
Title: Effect of Trumenba on Gonococcal Infections in Adolescents and Young Adults in the United States: A Retrospective Cohort Study
Brief Title: A Study to Learn About How Trumenba Vaccine Shots Work Against Gonorrhea Infection in Teenagers and Young Adults in the United States.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1971066; NCT05873751 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-05-15; First posted 2023-05-24 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Gonorrhea; Chlamydia; Meningococcal Vaccines
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections | interventions — MenB-FHbp vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Trumenba +MenACWY Vaccinated: Exposure Cohort that received at least one dose of Trumenba and MenACWY vaccine
  Interventions: Biological: Trumenba Vaccine; Biological: MenACWY Vaccine
- MenACWY Only Vaccinated: Non-exposure (reference cohort) that received at least one dose of MenACWY vaccine and no Trumenba vaccine.
  Interventions: Biological: MenACWY Vaccine

INTERVENTIONS:
Biological: Trumenba Vaccine — Trumenba vaccine given as standard of care
  Groups: Trumenba +MenACWY Vaccinated
Biological: MenACWY Vaccine — MenACWY Vaccine given as standard of care

SUMMARY:
Brief Summary:

The main purpose of the study is to learn about how well Trumenba vaccine shot works against gonorrhea infection.

This study looks at data records from a database in the United States.

This study includes patient's data from the database who:

* Are 15-30 years old.
* Have received at least one dose of Trumenba and a MenACWY vaccine or who have received only MenACWY vaccine.

This data has already been collected in the past and is being studied between April and June of 2023.

DETAILED DESCRIPTION:
This study is a retrospective cohort study including individuals registered and available in the PharMetrics Plus database from 01 Jan 2016 to 31 Dec 2022 In order to estimate the effect of Trumenba vaccination, the cumulative incidence rate over time of the defined disease of interest among Trumenba + MenACWY vaccines will be compared to that among MenACWY vaccinees. Stratified analysis will be made by age groups, gender and state of residence

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of 15-30 years old registered in the PharMetrics Plus system
2. Individuals having the index vaccination event at the age of 15-30 in 2016-2021

Exclusion Criteria:

1. Individuals having any dose of Bexsero at any time during the study period and prior to the study
2. Individuals with incomplete information on variables to be collected.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female adolescents and young adults 15-30 years old included in the PharMetrics claims database from 01Jan2016 through 31Dec2022 Individuals in this cohort who have received the index vaccination between 2016 and 2021.
Sampling Method: Non-Probability Sample
Enrollment: 1307378 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1971066

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (15-30 years of age) who received at least one dose of Trumenba and at least one dose of MenACWY prior to their Trumenba vaccination, between 01 January 2016 and 31 December 2021, were identified and their data (01 January 2016 to 31 December 2022) was retrieved from "IQVIA PharMetrics Plus" database. Available retrospective data was evaluated per objectives of the study during approximately 11 months.
Groups:
- Exposed Cohort: Vaccinated With Trumenba + MenACWY: Participants who had received at least one dose of Trumenba and at least one dose of MenACWY vaccine (prior to the Trumenba vaccination) between 01 January 2016 to 31 December 2021, their data was included in this retrospective study. Vaccination was not administered under this study.
- Non-Exposed Cohort: Vaccinated With MenACWY Only: Participants who had received at least one dose of MenACWY (but no doses of Trumenba vaccine) between 01-January-2016 to 31-December-2021, their data was included in this retrospective study. It is a reference cohort for this study. Vaccination was not administered under this study.
Period: Overall Study
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only
Started | 214552 | 1092826
Completed | 214552 | 1092826
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants whose data were included in this retrospective study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only | Total
Number analyzed (Participants) | 214552 | 1092826 | 1307378
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.97 (1.32) | 17.18 (1.99) | 17.15 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109013 | 553213 | 662226
  Male | 105539 | 539613 | 645152
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Northeast | 36193 | 199905 | 236098
  United States: South | 85947 | 390076 | 476023
  United States: Midwest | 68134 | 334106 | 402240
  United States: West | 23963 | 161031 | 184994
  United States: Unknown | 315 | 7708 | 8023

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Gonococcal Infection After at Least 1 Dose of Trumenba to Determine Vaccine Effectiveness (VE)
Description: Number of participants (cases) with infection of interest were reported. If a participant had repeated infection only first occurrence was considered, hence one participant with infection was counted only once. VE was calculated as 1 minus the hazard ratio (HR) multiplied by 100. VE is reported as part of statistical data in this outcome measure. The index date (zero time) was the date of the last dose of Trumenba vaccination, after at least one dose of MenACWY for the exposed cohort and first date of MenACWY vaccination for the unexposed cohort.
Time Frame: During follow-up of maximum of 83.5 months (from 14 days after the index date up to 31 December 2022; available retrospective data evaluated for approximately 11 months of this study)
Population: All eligible participants whose data were included in this retrospective study.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only
Number analyzed (Participants) | 214552 | 1092826
Participants | 316 | 2327
Statistical Analysis 1: Comparison: Exposed Cohort: Vaccinated With Trumenba + MenACWY vs Non-Exposed Cohort: Vaccinated With MenACWY Only; Test type: Other; Calibrated VE = 2.74, 95% CI 2-sided [-10.35 to 15.59] — VE = 1 - HR*100. The HRs were estimated by exponentiating the coefficient for the vaccine variable in the model. VE was adjusted for the covariates age, gender, and US census region

2. Secondary Outcome: Number of Participants With Gonococcal Infection After at Least 2 Doses of Trumenba to Determine VE
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All eligible participants whose data were included in this retrospective study. "Overall Number of Participants Analyzed" signifies participants who received at least two doses of Trumenba were included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only
Number analyzed (Participants) | 92661 | 1092826
Participants | 165 | 2327
Statistical Analysis 1: Comparison: Exposed Cohort: Vaccinated With Trumenba + MenACWY vs Non-Exposed Cohort: Vaccinated With MenACWY Only; Test type: Other; Calibrated VE = -2.2, 95% CI 2-sided [-23.50 to 13.85] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Chlamydial Infection After at Least 1 Dose of Trumenba to Determine VE
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All eligible participants whose data were included in this retrospective study.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only
Number analyzed (Participants) | 214552 | 1092826
Participants | 1138 | 7261
Statistical Analysis 1: Comparison: Exposed Cohort: Vaccinated With Trumenba + MenACWY vs Non-Exposed Cohort: Vaccinated With MenACWY Only; Test type: Other; Calibrated VE = 2.74, 95% CI 2-sided [-10.35 to 15.59] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Chlamydial Infection After at Least 2 Doses of Trumenba to Determine VE
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only
Number analyzed (Participants) | 92661 | 1092826
Participants | 584 | 7261
Statistical Analysis 1: Comparison: Exposed Cohort: Vaccinated With Trumenba + MenACWY vs Non-Exposed Cohort: Vaccinated With MenACWY Only; Test type: Other; Calibrated VE = -2.2, 95% CI 2-sided [-23.50 to 13.85] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Data for adverse events and deaths were not assessed/evaluated during the study; hence timeframe is not applicable.
Description: This study involved data that existed as structured data and in these data sources individual identifying information was not available. The minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) could not be met. Hence, adverse events were not planned to be evaluated.
Arm/Group | Exposed Cohort: Vaccinated With Trumenba + MenACWY | Non-Exposed Cohort: Vaccinated With MenACWY Only
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT05873751/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/51/NCT05873751/SAP_001.pdf